CLINICAL TRIAL: NCT02829684
Title: Implementation of a National Register of Children and Adults Presenting Prader-Willi Syndrome
Brief Title: Register of Patients With Prader-Willi Syndrome
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 07 315 03
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Data collection — This register will follow the evolution of the clinical practices and their consequences in the health of the patients, in all regions of France in order to have a national register. for Children and adults.

SUMMARY:
Prader-Willi Syndrome (PWS) is a rare syndrome with a prevalence of 15 to 20 000 at birth. PWS represents a large fraction of mental retardation syndromes due to a genetic cause and the most frequent cause of genetic obesity. The majority of the patients are seen by paediatricians. This syndrome is responsible for severe physical, psychological and social impairments.

The diversity and the severity of the manifestations of this disease explain the requirement of multidisciplinary care which deserve specific evaluation. Today the follow-up and management of a great proportion of these patients are greatly insufficient if not absent.

Teams strongly lack information on the natural history of this severe disease and on the factors involved in its evolution and the outcome of these patients throughout life. The present project is to implement a register in the whole country for children and adult patients

ELIGIBILITY:
Inclusion Criteria:

* all subjects with a Prader-Willi Syndrome

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be included by the paediatric endocrinologists or the endocrinologists for adults of each region based on their own recruitment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
collect data about patients | Baseline
  Circumstances of diagnosis, genetic diagnosis, modalities of follow-up and clinical management and a questionnaire to evaluate quality of life of the family and social data

SECONDARY OUTCOMES:
collect data about patients | During 10 years at least
  modalities of follow-up and clinical management and a questionnaire to evaluate quality of life of the family and social data

CONTACTS AND LOCATIONS:
Overall Officials: Tauber Maité, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Children, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pacoricona Alfaro DL, Lemoine P, Ehlinger V, Molinas C, Diene G, Valette M, Pinto G, Coupaye M, Poitou-Bernert C, Thuilleaux D, Arnaud C, Tauber M. Causes of death in Prader-Willi syndrome: lessons from 11 years' experience of a national reference center. Orphanet J Rare Dis. 2019 Nov 4;14(1):238. doi: 10.1186/s13023-019-1214-2. PMID 31684997